CLINICAL TRIAL: NCT02898181
Title: Low Level Transcutaneous Tragus Stimulation to Reduce Inflammation, Dyspnea and Improve Heart Rate Variability in Acute Decompensated Heart Failure
Brief Title: Low Level Tragus Stimulation in Acute Decompensated Heart Failure
Acronym: TREAT-HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6778
Record Dates: First submitted 2016-09-01; First posted 2016-09-13 (Estimated); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Acute Decompensated Heart Failure
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Tragus Stimulation (Experimental): In this group patients will receive neuromodulation for 2 hours daily
  Interventions: Device: Neuromodulation
- Control group (No Intervention): Sham neuromodulation will be done

INTERVENTIONS:
Device: Neuromodulation — Active LLTS will be performed by use of a transcutaneous electrical nerve stimulation Parasym neuromodulation system with electrodes attached to the ear. Neuromodulation will be applied continuously for 2 hours daily.
  Arms: Tragus Stimulation

SUMMARY:
Acute Decompensated Heart Failure (ADHF) is a major cause of morbidity and mortality. It is associated with increased systemic inflammation. Previous studies have demonstrated increased levels of cytokines such as C-reactive protein (CRP), interleukin-1 (IL-1), interleukin-6 (IL-6), interleukin-10 (IL-10) and Tumor Necrosis Factor alpha (TNFα) in patients with heart failure (HF). Increased activity of sympathetic nervous system in ADHF is linked to inflammation. Previous anti-inflammatory drug therapies in HF have demonstrated no significant impact on cardiovascular outcomes. Low-level vagus nerve stimulation (LLVNS) is a non-invasive way to modulate autonomic tone and thereby inflammation. Vagal nerve stimulation is thought to increase the parasympathetic activity and suppress the sympathetic activity. Clinical studies of vagal stimulation in chronic HF have been negative. Recent experimental and clinical data suggest that low level tragus nerve stimulation (LLTNS) may produce the same desired neuromodulator effect compared to LLVNS. It is however unknown if LLTNS in ADHF will directly lead to a reduction in the levels of pro-inflammatory cytokines (CRP, IL-1, IL-6 and TNF-α) and an increase in the level of anti-inflammatory marker IL-10. heart rate variability may also be abnormal in ADHF. The objective of this proposal is to determine the impact of LLTS on inflammatory cytokines, heart failure biomarkers(Pro BNP) and HRV in patients with ADHF.In addition we will study the impact on dyspnea resolution and change in renal function during hospitalization.

Patients will be randomized to either active or sham stimulation (2 hours daily). Serum collected will (post-admission and discharge day) will be used for cytokine measurement. We will also measure daily ECG to assess HRV and patient assessed dyspnea scale.This investigation will likely establish the first evidence of the effects of LLTS on the suppression of inflammation and improvement in dyspnea, natriuretic peptides, renal function and HRV in patients presenting with ADHF.

DETAILED DESCRIPTION:
Acute Decompensated Heart Failure (ADHF) is a major cause of morbidity and mortality. It is associated with increased systemic inflammation and poor outcomes.

Previous studies have demonstrated increased inflammation in patients with heart failure (HF). Increased activity of sympathetic nervous system in ADHF is linked to inflammation. Previous anti-inflammatory drug therapies in HF have demonstrated no significant impact on cardiovascular outcomes.

Low-level vagus nerve stimulation via stimulation of teh Tragus (LLTS) is a non-invasive way to modulate autonomic tone and thereby inflammation. Vagal nerve stimulation is thought to increase the parasympathetic activity and suppress the sympathetic activity. Recent experimental and clinical data suggest that low level tragus nerve stimulation (LLTS) may produce the same desired neuromodulator effect compared to LLVNS.

It is however unknown if LLTS in ADHF will directly lead to sympathetic tone reduction and increase in parasympathetic tone, or neuromodulation and lead to reduction in the levels of pro-inflammatory cytokines (CRP, IL-1, IL-6 and TNF-α) and an increase in the level of anti-inflammatory marker IL-10.

Autonomic tone could be assessed using heart rate variability. The objective of this proposal is to determine the impact of LLTS on inflammatory cytokines and HRV in patients with ADHF.

Patients will be randomized to either active or sham stimulation (2 hours daily).

Serum collected will (post admission and discharge day) will be used for cytokine and biomarker measurement. We will also measure 10-15 minute ECG to assess HRV. Dyspnea will be determined using patient assessment tool(visual analog scale).This investigation will likely establish the first evidence of effects of LLTS on suppression of inflammation and improvement in dyspnea scale, renal function and HRV in patients presenting with ADHF.

ELIGIBILITY:
Inclusion Criteria:

Patients admitted with ADHF

Exclusion Criteria:

1. Refusal to consent
2. Complex congenital heart disease (Tetralogy of Fallot patients, single ventricle physiology)
3. Recurrent vaso-vagal syncopal episodes
4. Unilateral or bilateral vagotomy
5. Sick sinus syndrome
6. 2nd or 3rd degree AV block
7. bifascicular block or prolonged 1st degree AV block (PR>300ms)
8. Pregnant patients
9. Prisoners
10. Advanced renal dysfunction(defined as eGFR < 30, stage 4 or 5 chronic kidney disease)
11. Hepatitis C or HIV
12. Acute Myocardial infarction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-09; Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Change in Interleukin (IL) levels | From admission to discharge- over average 3-6 days
  Interleukin level
Change in TNF-alpha levels | From admission to discharge- over average 3-6 days
  TNF level
Change in CRP levels | From admission to discharge- over average 3-6 days
  CRP level
Change in Pro BNP and renal function(creatinine) levels | From admission to discharge- over average 3-6 days
  Pro BNP level

SECONDARY OUTCOMES:
Change in HRV | From admission to discharge- over average 3-6 days
  Heart rate variability measures such time and frequency domains

OTHER OUTCOMES:
Change in level of dyspnea | From admission to discharge- over average 3-6 days
  Dyspnea will be determined using simple tool called visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Dasari, MD,MPH, Principal Investigator — OUHSC
Locations (1):
- OUHSC, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dasari TW, Chakraborty P, Mukli P, Akhtar K, Yabluchanskiy A, Cunningham MW, Csiszar A, Po SS. Noninvasive low-level tragus stimulation attenuates inflammation and oxidative stress in acute heart failure. Clin Auton Res. 2023 Dec;33(6):767-775. doi: 10.1007/s10286-023-00997-z. Epub 2023 Nov 9. PMID 37943335
- [Derived] Dasari T, Chakraborty P, Mukli P, Akhtar K, Yabluchanskiy A, Cunningham MW, Csiszar A, Po SS. Noninvasive low-level tragus stimulation attenuates inflammation and oxidative stress in acute heart failure. Res Sq [Preprint]. 2023 Sep 11:rs.3.rs-3323086. doi: 10.21203/rs.3.rs-3323086/v1. PMID 37790298